CLINICAL TRIAL: NCT01296958
Title: Targeted Screening for Taenia Solium Tapeworms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: National University of San Marcos, Peru (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Seth E O'Neal, MD MPH, Assistant professor, Oregon Health and Science University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 1R21NS069275-01 (NIH); 1R21NS069275-01 (NIH)
Record Dates: First submitted 2011-02-15; First posted 2011-02-16 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Taenia Solium Taeniasis
Keywords: Taenia solium; cysticercosis; neurocysticercosis
MeSH Terms: conditions — Taeniasis; Cysticercosis; Neurocysticercosis | interventions — Niclosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Targeted screening (Experimental): Screening for intestinal tapeworm carrier followed by treatment with niclosamide as indicated.
  Interventions: Drug: Niclosamide
- Education (Active Comparator): Community education about Taenia solium prevention.
  Interventions: Behavioral: Community education campaign

INTERVENTIONS:
Drug: Niclosamide — Single oral dose of niclosamide determined by weight (dose: 11 to 34kg receive 1 gram, 35 to 50kg receive 1.5 grams, over 50kg receive 2 grams)
  Arms: Targeted screening
Behavioral: Community education campaign — Education about prevention of Taenia solium infection provided in a single short (20 minute) interaction with the participant. Education was verbal with visual aids.
  Arms: Education

SUMMARY:
The purpose of this study is to determine whether screening and treatment of tapeworm carriers can decrease community transmission of Taenia solium parasitic infection.

ELIGIBILITY:
Inclusion Criteria:

* All community members are eligible

Exclusion Criteria:

* Inability to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1811 (Actual)
Dates: Start 2011-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Porcine seroprevalence | Every 4 months

SECONDARY OUTCOMES:
Intestinal tapeworm prevalence | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Seth E ONeal, MD MPH, Principal Investigator — Oregon Health and Science University; Armando Gonzalez, DVM PhD, Principal Investigator — San Marcos University School of Veterinary Medicine
Locations (1):
- San Marcos University, Lima, Peru